CLINICAL TRIAL: NCT04148690
Title: Assessing the Impact of IPTp Uptake Among Pregnant Women Attending Antenatal Clinic and Feasibility of Malaria Surveillance to Community Based Surveillance in Tanzania
Brief Title: Assessing the Impact of Group Antenatal Care on IPTp Uptake in Tanzania
Acronym: GANC-TZ
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Group intervention suspended due to COVID-19 risk
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Jhpiego (Other); Ministry of Health, Tanzania (Other Government)
Responsible Party: Principal Investigator, Julie Gutman, Medical Officer, Strategic and Applied Science Unit, Malaria Branch, Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 7226 GANC-TZ
Record Dates: First submitted 2019-10-25; First posted 2019-11-01 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Malaria; Malaria in Pregnancy
Keywords: Group antenatal care; Surveillance; Tanzania; Malaria in Pregnancy
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: This will be a cluster randomized controlled trial conducted over an 18-month period. Facilities will be randomized 1:1 to control and intervention arms.
Who Masked: Outcomes Assessor
Masking Description: the outcomes will be assessed through conduct of a cross sectional survey; those conducting the survey will not be informed as to which arm the women were in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ANC Intervention (Experimental): Clinics in the group ANC intervention arm offer group Antenatal Care to women who present for their initial visit prior to 24 weeks provided that they intend to remain in the area for the duration of the pregnancy, and agree to participate in GANC. Women not enrolled in group ANC will receive standard ANC per ministry of health protocols.
  Interventions: Other: Group antenatal care (GANC)
- Routine ANC (Active Comparator): Clinics will offer only standard ANC per ministry of health protocols.
  Interventions: Other: Standard antenatal care

INTERVENTIONS:
Other: Group antenatal care (GANC) — Group antenatal care (GANC) is a service delivery model where women with pregnancies of similar gestational age are brought together for antenatal care (ANC), incorporating information sharing and peer support.
  Arms: Group ANC Intervention
Other: Standard antenatal care — Routine antenatal care as recommended by th Ministry of Health of Tanzania
  Arms: Routine ANC

SUMMARY:
Group antenatal care (GANC) is a service delivery model where women with pregnancies of similar gestational age are brought together for antenatal care (ANC), incorporating information sharing and peer support. This model provides selected aspects of clinical care to women in the group at the same time during group visits, as well as creating a support group of women at a similar stage in pregnancy, to improve the quality of care and engagement of women in the ANC process, ultimately leading to better retention in care. Initial studies have suggested that this improves uptake of intermittent preventive treatment in pregnancy (IPTp) among women who participate, but have not evaluated the effect at community level. The investigators propose to assess whether use of the GANC model in Tanzania can improve the quality of ANC as compared to standard individual ANC, by measuring uptake of recommended interventions, primarily IPTp.

Recent data from Tanzania and Kenya suggest that malaria parasitemia prevalence among pregnant women correlates with the prevalence among children under five, and could be used to track trends over time.3-5 The very high coverage of ANC (>80% attending at least one ANC contact), suggests that pregnant women could be a good sentinel population that could be readily tracked over time. However, pregnant women represent only about 5% of the overall population, thus, it is important to demonstrate that the trends in malaria prevalence and household level coverage of interventions reported by pregnant women attending ANC is representative of coverage among the general population. If validated, these data could be used to augment or even replace the data on coverage of interventions collected through the use of malaria indicator surveys, which are expensive and infrequently conducted, and generally only powered to the regional level.

DETAILED DESCRIPTION:
Project Background Group antenatal care (GANC) is a service delivery model where women with pregnancies of similar gestational age are brought together for antenatal care (ANC), incorporating information sharing and peer support. This model provides selected aspects of clinical care to women in the group at the same time during group visits, as well as creating a support group of women at a similar stage in pregnancy, to improve the quality of care and engagement of women in the ANC process, ultimately leading to better retention in care. Initial studies have suggested that this improves uptake of intermittent preventive treatment in pregnancy (IPTp) among women who participate, but have not evaluated the effect at community level. The investigators propose to assess whether use of the GANC model in Tanzania can improve the quality of ANC as compared to standard individual ANC, by measuring uptake of recommended interventions, primarily IPTp. Tanzania have been selected as coverage of early ANC is high, with 98% of women receiving ANC from a trained provider in Tanzania and 83% in Benin,1 with a median age of initiation of five and four months, respectively. Coverage of 4 ANC visits, however, is sub-optimal: just 36% in Geita region of Tanzania. Despite the relatively early initiation of ANC, in Tanzania only 56% and 26% of women received two and three doses of IPTp.

Recent data from Tanzania and Kenya suggest that malaria parasitemia prevalence among pregnant women correlates with the prevalence among children under five, and could be used to track trends over time.3-5 The very high coverage of ANC (>80% attending at least one ANC contact), suggests that pregnant women could be a good sentinel population that could be readily tracked over time. However, pregnant women represent only about 5% of the overall population, thus, it is important to demonstrate that the trends in malaria prevalence and household level coverage of interventions reported by pregnant women attending ANC is representative of coverage among the general population. If validated, these data could be used to augment or even replace the data on coverage of interventions collected through the use of malaria indicator surveys, which are expensive and infrequently conducted, and generally only powered to the regional level.

Study Aims

Primary Objectives:

1. GANC: Assess whether GANC is associated with to improved uptake of IPTp; specifically, to assess whether the proportion of pregnant women receiving 3 or more doses of IPTp is higher in the catchment areas of facilities implementing the GANC intervention as compared to the catchment areas of control facilities without GANC.
2. ANC data for surveillance: Pilot data collection from women at 1st ANC and validate whether the results obtained from this population are representative of the population as a whole.

Secondary Objectives:

GANC

1. To assess whether implementation of GANC is associated with to a greater proportion of women completing the recommended number of ANC visits compared to control facilities without GANC.
2. To assess whether the implementation of GANC leads to earlier initiation of ANC compared to control facilities without GANC, as women can only participate in GANC if they present <24 weeks.
3. To assess whether GANC is associated with increased utilization of facility-based delivery
4. To assess whether GANC is associated with improved quality of care (defined as the coverage of key ANC interventions- blood pressure, urine test, blood test, tetanus, iron-folic acid (IFA), albendazole, insecticide treated bednet (ITN), IPTp)
5. To assess the feasibility and acceptability of increasing the coverage of GANC
6. To assess the costs and cost effectiveness of GANC versus individual ANC (standard of care)

   ANC data for Surveillance
7. To understand the acceptability to pregnant women and healthcare workers of being asked/asking these additional questions during ANC contacts.
8. To quantify the time per woman required to collect data on coverage of malaria control interventions into ANC
9. To assess the correlation between the prevalence of malaria by rapid diagnostic test (RDT) among pregnant women attending 1st ANC and among children under 5 measured in cross sectional household surveys
10. To explore optimal data collection strategies and determine how best to operationalize them (i.e., should data be collected and recorded by ANC providers or another cadre; e.g., a community health worker stationed at the clinic).

Methodology Study design: This will be a cluster randomized controlled trial conducted over an 18-month period. Facilities will be randomized 1:1 to control and intervention arms. In the control arm, ANC care will be delivered as per standard practice. In the intervention sites, women presenting for first ANC prior to 24 weeks will be offered the opportunity to join group care (as long as there is still space in an appropriate group) starting with the 2nd visit; women presenting after 24 weeks or declining to join a group will receive standard ANC care.

Baseline and end line cross sectional household surveys will be conducted 18 months apart to measure the proportion of women living in the facility catchment areas who have completed a pregnancy (ie. given birth) within the past 12 months in each community who received 1, 2, 3, 4, and 5+ doses of IPTp, the timing of initiation of ANC, number of total ANC visits, facility-based delivery, birth outcomes, as well as validate the representativeness of data on parasite prevalence, insecticide treated net (ITN) ownership and use, and care seeking. The sample size in each country will be sufficient to allow for an estimate of the effect of GANC for each country, as the effectiveness of this model is dependent on the proportion of women who attend ANC early, which is somewhat higher in Benin than in Tanzania.

Implications The results will be used by the Ministries of Health (MOH) in Tanzania to decide: whether to expand the use of GANC as a strategy to improve quality of care and increase utilization of ANC; and whether pregnant women attending first ANC can be used as a sentinel population to improve surveillance of malaria control interventions.

Expected findings and dissemination The investigators will share the results of this study with the MoHs and the partners working in malaria and maternal and child health through: country-based technical working groups in malaria and maternal and newborn health; community leaders; and women's associations-as well as dissemination events and print materials. The findings will contribute to the evidence to determine whether GANC is associated with improved ANC attendance, IPTp uptake, and quality of care (as defined as the delivery of specific interventions), and whether it should be scaled-up in other suitable malaria endemic regions. The findings on ANC surveillance will contribute to the evidence about whether this method of surveillance is effective and should be scaled up. The results will also be presented in both local and international scientific meetings and published in a peer-reviewed journal.

ELIGIBILITY:
Pregnant women for GANC and ANC surveillance:

Inclusion Criteria

* Pregnant women residing in the facility catchment area, who present for initial ANC visit prior to 24 weeks are eligible to participate in GANC provided that they intend to remain in the area for the duration of the pregnancy, and agree to participate in GANC. All women attending first ANC at participating facilities will be asked to respond to a short list of questions regarding the coverage of malaria control interventions in their household.

Exclusion criteria

• Pregnant women: Women will be excluded from participation in GANC if they initiate ANC care >24 weeks gestation, if there are no available groups that they can join, if they do not intend to remain in the facility catchment area for the duration of the study, or if they are not available during the times the group intends to meet. Women will also be excluded if they do not speak Swahili, as group discussions will be conducted in Swahili.

Recently pregnant women (for cross sectional household surveys) Inclusion Criteria • To be included in the women's question portion of the baseline and end line household (HH) surveys, women must be between the ages of 15-49 years, have been pregnant/delivered in the previous 12 months, consent to participation, and will be eligible for inclusion in surveys regardless of where the woman gave birth (i.e., whether at home or in facility). All pregnant/recently pregnant women will be included in the cross sectional survey, but the sample size is calculated in order to identify those who have completed pregnancies in the past 12 months. There will be a short subset of demographic and knowledge questions which will be asked of all households (either female or male respondents) during the baseline and end line surveys, regardless of whether there are any recently pregnant women in the household.

Exclusion criteria • Women who gave birth in the past 12 months, but are <15 or >49 years will be excluded. Those who last delivered a child over twelve months ago will be excluded from survey questions specific to recently pregnant women, but may answer questions related to community perception or general demographics. For qualitative research, the same criteria will be used.

Children (for blood sampling during the cross sectional household surveys) Inclusion Criteria

• Children between the ages of 6-59 months will be included provided that they are living in households interviewed during the baseline or end line cross sectional survey and a parent or legal guardian provides consent for their participation

Exclusion criteria • Children will be excluded if they are <6 months or >59 months, or if their parent/guardian is not present or does not provide consent

Providers:

Inclusion Criteria

* ANC provider who has had at least six months of work experience
* Health facility in-charge
* Health management information system (HMIS) focal person

Exclusion criteria

• Those who have been working in the health facility for less than six months will not be interviewed due to low levels of relevant experience or exposure to the intervention.

Policy makers:

Inclusion Criteria

• In depth interviews may be conducted with program managers (malaria, reproductive health, and statistics/ data collection officers) at the district, regional and national levels

Exclusion criteria

• None

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4515 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Change in proportion of recently pregnant women receiving IPTp3 | Change between 0 and 18 months of implementation
  Proportion of recently pregnant women receiving IPTp3 as measured by cross sectional household surveys
Correlation between ANC data and population data | Through study completion, an average of 1 year
  Correlation between ANC data and population data collected during cross sectional survey on ITN ownership and care seeking behavior among children

SECONDARY OUTCOMES:
Change in ANC coverage | Change between 0 and 18 months of implementation
  Proportion of recently pregnant women completing the four, six, and eight ANC visits as measured by cross sectional household survey
Change in Gestational age at initiation of ANC | Change between 0 and 18 months of implementation
  Mean gestational age at initiation of ANC measured by cross sectional household survey
Change in Proportion of women who recently gave birth who received blood pressure, urine test, blood test, tetanus, IFA, albendazole, ITN, and IPTp | Change between 0 and 18 months of implementation
  Change in Proportion of women who recently gave birth who received blood pressure, urine test, blood test, tetanus, IFA, albendazole, ITN, and IPTp as measured by cross sectional household surveys
Change in Proportion of women who recently gave birth who had a facility-based delivery as measured by cross sectional household surveys | Change between 0 and 18 months of implementation
Prevalence of malaria by RDT among pregnant women attending 1st ANC | throughout study period; average of once per month
Prevalence of malaria by RDT among among children under 5 | throughout study period; average of once per year
Difference in provider time required to deliver GANC versus individual ANC | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Lemwayi, MD, Principal Investigator — Jhpiego; Julie R Gutman, MD MSc, Principal Investigator — Centers for Disease Control and Prevention; Mary Drake, Principal Investigator — Jhpiego
Locations (1):
- Chato District Hospital, Chato, Tanzania

IPD SHARING:
Plan to Share IPD: No
Individual participant data may only be made available upon specific request after appropriate approvals for data sharing have been granted by Tanzanian authorities